CLINICAL TRIAL: NCT04457492
Title: Applying Functional Electrical Stimulation to Facial Muscles After Acute Paralysis
Brief Title: Functional Electrical Stimulation for Facial Muscles
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI Relocation
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-5743
Record Dates: First submitted 2020-06-08; First posted 2020-07-07 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Facial Nerve Paresis
Keywords: Facial Nerve Paralysis; Functional Electrical Stimulation; Rehabilitation
MeSH Terms: conditions — Bell Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acute Facial Nerve Injury with Intact Facial Nerve (Experimental): 40 sessions of FES (in a 14 week period)
  Assessments will be taken during the beginning, middle, and end of each study arm.
  Interventions: Other: Application of FES to the Face
- Facial Nerve Grafting After Surgical Excision (Experimental): 40 sessions of FES (in a 14 week period)
  Assessments will be taken during the beginning, middle, and end of each study arm.
  Interventions: Other: Application of FES to the Face
- Standard of Care Group (No Intervention): No FES
  Assessments will be taken at the same intervals as the interventions group.

INTERVENTIONS:
Other: Application of FES to the Face — Functional electrical stimulation (FES) for facial paralysis is a technique in which muscles are electrically stimulated.
  Arms: Acute Facial Nerve Injury with Intact Facial Nerve; Facial Nerve Grafting After Surgical Excision

SUMMARY:
Partial or complete facial paralysis is the weakness of muscles of facial expression. Facial paralysis causes physical, social and emotional problems. Functional electrical stimulation (FES) for facial paralysis is a technique in which muscles are electrically stimulated, causing them to contract This study is designed to help patients with facial nerve weakness.

ELIGIBILITY:
Inclusion Criteria:

* Patients experiencing unilateral facial nerve paralysis Brackmann 5/6 or 6/6.

Exclusion Criteria:

* History of epilepsy or seizures.
* Individuals with metal orthopedic implants in the mouth (e.g. plates or screws).
* Individuals suffering from fibromyalgia.
* Individuals currently receiving any form of transcranial brain stimulation (e.g. rTMS, ECT, or MST).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Change in Lagophthalmos Over 14 weeks | Measured at week 0, 7 and 14
  Change in ability to close eyelids, measured in mm
Change in Elevation of Corner of Mouth Over 14 weeks | Measured at week 0, 7 and 14
  Change in ability to raise corner of mouth, measured in mm
Change House-Brackmann Scale Measurement Over 14 weeks | Measured at week 0, 7 and 14
  The House-Brackmann facial nerve grading scale is a measure of facial nerve impairment. The scale ranges from values 1 to 6, with larger values indicating greater facial nerve impairment.
FaCE Questionnaire | Administered at week 0, 7 and 14
  Patient-based instrument to measure both facial impairment and disability. This will be used to identify patient's perceived change in facial impairment for the duration of the study period.
Change in Facial Movements Over 14 weeks | Measured at week 0, 7 and 14
  A video will be taken of the patient undergoing standard facial movements
Study Interview | Administered at week 0, 7 and 14
  A structured interview questionnaire administered by a study team member to identify any changes to the therapy that may be needed before further studies are conducted

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Chepeha, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada